CLINICAL TRIAL: NCT07163897
Title: Validation of a Portable Ankle Arthrometer
Status: Not yet recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jay Hertel, PhD, ATC, Joe H. Gieck Professor of Sports Medicine; Chair of the Department of Kinesiology; Licensed Athletic Trainer, University of Virginia
Other Study IDs: 302715
Record Dates: First submitted 2025-08-20; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Chronic Ankle Instability, CAI; Ankle Sprain; Healthy
Keywords: Arthrometer; Ankle; Validity; Reliability
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy: Individuals that have never sprained their ankle.
  Interventions: Device: Cobra Ankle Arthrometer
- Copers: Individuals that have sprained their ankle one time, with no residual problems.
  Interventions: Device: Cobra Ankle Arthrometer
- CAI: Individuals that have been diagnosed with chronic ankle instability.
  Interventions: Device: Cobra Ankle Arthrometer
- Acute Sprain: Individuals that have sprained their ankle in the last 96 hours.
  Interventions: Device: Cobra Ankle Arthrometer

INTERVENTIONS:
Device: Cobra Ankle Arthrometer — This is a prototype portable ankle arthrometer designed to measure the laxity of the ankle joint.

SUMMARY:
The purpose of this study is to assess the validity and reliability of a prototype portable ankle arthrometer in various populations. There are two aims to this study. Aim 1 will look to determine the reliability and validity of a prototype portable ankle arthrometer on young adults with no history of ankle sprain, copers, and young adults with chronic ankle instability. It is hypothesized that the prototype portable ankle arthrometer will be a valid and reliable tool to assess joint laxity across the three different populations. Aim 2 will look to determine the validity of a prototype portable ankle arthrometer in young adults with an acute ankle sprain across multiple timepoints in their first month post injury. It is hypothesized that the prototype portable ankle arthrometer will be a valid tool to assess joint laxity at three different timepoints for the same individual.

DETAILED DESCRIPTION:
Aim 1: Participants will report to the Exercise and Sport Injury laboratory to provide informed consent before any study procedures take place. Following consent, there will be an approximate 1 hour data collection period. There will be 2 different days of data collection, with informed consent being provided only at the first session.

Demographics & Health History: Participants will answer several surveys including a medical history questionnaire, physical activity readiness questionnaire (ParQ), international physical activity questionnaire (IPAQ - short form), identification of functional ankle instability (IdFAI), and a foot and ankle ability measure (FAAM). Measures of age, height, weight, sex, and race or ethnicity will be recorded by practitioners prior to testing. Information gathered will be used to ensure all participants fit the study inclusion criteria.

Instrumentation will include a prototype portable ankle arthrometer created by Luna Labs to measure joint laxity and a GE Healthcare Ultrasound Machine to also measure joint laxity.

Participants will first undergo a series of physical examination tests performed by a Licensed Athletic Trainer. Participants will remain seated on the exam table, and the study team member will perform the "Anterior Drawer Test of the Ankle" and the "Talar Tilt Test" to assess the stability of the participants ankle ligaments.

Following the physical exam tests, participants will remain seated on the exam table and will be outfitted with the ankle arthrometer. Once the arthrometer is fitted, participants will have their foot placed in various positions, and the arthrometer will record measures.

Following the ankle arthrometer, participants will remain seated on the exam table and the ultrasound imaging unit will be used to assess joint laxity in the same positions that were used for the ankle arthrometer.

Following the completion of ultrasound images, participants will be dismissed. Participants will then report back a week later for visit 2. Visit 2 consist of the physical exam tests, ankle arthrometer, and ultrasound imaging again.

Following visit 2, participation in the study will be complete.

Aim 2: Participants will report to the Exercise and Sport Injury laboratory to provide informed consent before any study procedures take place. Following consent, there will be an approximate 1 hour data collection period. There will be 3 different days of data collection, with informed consent being provided only at the first session.

Demographics & Health History: Participants will answer several surveys including a medical history questionnaire, physical activity readiness questionnaire (ParQ), international physical activity questionnaire (IPAQ - short form), and a foot and ankle ability measure (FAAM). Measures of age, height, weight, sex, and race or ethnicity will be recorded by practitioners prior to testing. Information gathered will be used to ensure all participants fit the study inclusion criteria.

Instrumentation will include a prototype portable ankle arthrometer created by Luna Labs to measure joint laxity and a GE Healthcare Ultrasound Machine to also measure joint laxity.

Participants will first undergo a series of physical examination tests performed by a Licensed Athletic Trainer. Participants will remain seated on the exam table, and the study team member will perform the "Anterior Drawer Test of the Ankle" and the "Talar Tilt Test" to assess the stability of the participants ankle ligaments.

Following the physical exam tests, participants will remain seated on the exam table and will be outfitted with the ankle arthrometer. Once the arthrometer is fitted, participants will have their foot placed in various positions, and the arthrometer will record measures.

Following the ankle arthrometer, participants will remain seated on the exam table and the ultrasound imaging unit will be used to assess joint laxity in the same positions that were used for the ankle arthrometer.

Following the completion of ultrasound images, participants will be dismissed. Participants will then report back 2 weeks later for visit 2. Visit 2 consist of completion of the FAAM, physical exam tests, ankle arthrometer, and ultrasound imaging again. Visit 3 will consist of the same study procedure, however the timepoint will be 4 weeks after visit 1.

Following visit 3, participation in the study will be complete.

ELIGIBILITY:
Aim 1:

Inclusion Criteria:

* Young adults between the ages of 18 and 40.
* Willingness and ability to comply with scheduled visits and study procedures.
* Fit one of the three groups: 1. Healthy - no history of ankle sprain, 2. Copers - one previous ankle sprain with no residual problems, 3. Chronic Ankle Instability.
* Ability to sign consent.

Aim 2:

Inclusion Criteria:

* Young adults between the ages of 18 and 40.
* Willingness and ability to comply with scheduled visits and study procedures.
* Acute ankle sprain within the last 48-96 hours.
* Ability to sign consent.

Aim 1:

Exclusion Criteria:

* Previous history of ankle fracture.
* Diagnosis of Ehlers-Danlos Syndrome

Aim 2:

Exclusion Criteria:

* Previous history of ankle fracture.
* Diagnosis of Ehlers-Danlos Syndrome.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Ankle laxity | Aim 1: From Day 1 to the end of study after Day 2 (One week after Day 1). Aim 2: From Day 1 to the end of study after Day 3 (Four weeks after Day 1).
  Measured with both the ankle arthrometer and ultrasound imaging. Both will report units of displacement.

CONTACTS AND LOCATIONS:
Locations (1):
- UVA Department of Student Health and Wellness, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No